CLINICAL TRIAL: NCT03373370
Title: Project to Accelerate the Diagnosis of TTR Amyloidosis by Use of Molecular Biology in First Intention
Brief Title: Early Diagnosis of TTR Amyloidosis by Use of Molecular Biology
Acronym: ADDITION
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 16007
Record Dates: First submitted 2017-12-11; First posted 2017-12-14 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Polyneuropathy; Diagnosis; Idiopathic Progressive Neuropathy
MeSH Terms: conditions — Polyneuropathies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral neuropathies are diseases that affect the nervous system outside the brain and spinal cord, their prevalence is 1% in the general population, the causes are extremely varied with more than 200 identified causes; the main ones are diabetes, excessive alcohol consumption and chemotherapy. They may be sometimes disabling but generally preserve autonomy.

Transthyretin amyloidosis is a rare multisystematic hereditary disease with autosomal dominant transmission. They present usually as a peripheral neuropathies (FAP). They are due to a point mutation of the transthyretin gene (chr 18q). FAP is secondary to endoneurial amyloid deposits and are characterized by a slowly progressive sensory, motor and autonomic. FAP is the most severe hereditary polyneuropathy of the adult are irreversible and fatal within 5 to 12 years from onset.

Most frequent mutation of TTR gene is located on the second exon; but more than 100 mutations have been reported.

Prevalence of FAP is 1 per 1 million inhabitants. They have been reported until 1990s' in four endemic areas North of Portugal, Sweden, Japan and Majorca. In these areas, diagnosis is facilitated because of the stereotypical presentation : a length-dependent polyneuropathy with predominant involvement of thermal and pain sensations and autonomic dysfunction, early onset in the third decade and a predominant Met30 TTR mutation. Positive family history is frequent 85% (one of the parents is affected). Diagnosis requires detection of TTR mutation by molecular biology (blood sample) and characterization of amyloid deposit on labial salivary gland biopsy.

DETAILED DESCRIPTION:
Study of the TTR gene by complete sequencing; search for amyloidogenic mutations of the TTR gene (according to the site http: // amyloidosismutations.com / mut-attr.php) in the laboratory of molecular biology of the CHU BICÊTRE (APHP) managed by Pr Anne Mantel.

Preselection of the cases to be tested among the cases of peripheral neuropathies of indetermined cause referred via the network Cornamyl of which the reference centers of the neuromuscular diseases are belonging .

Currently, FAP is a worldwide disease. Diagnosis of TTR-FAP is extremely difficult and usually delayed by 4 years in non endemic areas for many reasons :

* positive family history are lacking in 50% of cases (sporadic forms).
* incomplete ability of biopsies to characterize amyloid deposits.
* clinical presentation is varied and may mimick many types of rare peripheral neuropathies: CIDP, axonal idiopathic polyneuropathy, upper limb neuropathies, recurrent carpal tunnel syndrome after surgery, ataxic neuropathy, motor neuropathy.

Conversely to endemic areas, look for V30M mutation is not enough to exclude TTR-FAP, TTR gene sequencing is required.

With the help of the french network for FAP (Cornamyl), cases have been identified in 81/100 geographical departments, with a wide genetic heterogeneity (41 mutations reported) ; age of onset is late: 75% after 50 yo.

ELIGIBILITY:
The initial criteria before amendment

Inclusion Criteria:

* A. Adult (>50 years old)
* Chronic Peripheral neuropathies (progressing since 12 months),
* Peripheral neuropathies documentated by ENMG.

  1. Chronic polyneuropathy with dysautonomia (orthostatic hypotension) without diabetes
  2. Atypical CIDP (situations C, D (even with high protid content on CSF) & E as defined by the French group for study of CIDP).
  3. Disabling neuropathy (gait or balance disorder)
  4. Neuropathies with upper limb onset who underwent previously CTS surgery without success.
  5. SLA-like syndrome : areflexia with sensory alterations on ENMG. 6: Deterioration of SNAPs' amplitudes on NCS > 30% in less than6 months by the same NCS laboratory Mandatory : A+B+C one of 1 to 6

Exclusion criteria :

* Amyloid deposit characterized on biopsy
* Causes of chronic polyneuropathy : Diabetes mellitus, Chronic alcoholic intoxication
* CIDP responding to IVIg or corticosteroids (improvement by 1 point of ONLS).
* Neuropathy associated with monoclonal gammapathy and i) anti-MAG activity or ii) POEMS syndrome or) CANOMAD syndrome.
* Ataxic Neuropathy due to vitamine B12 deficiency
* Ataxic Neuropathy due to IgM anti-MAG,
* CANOMAD syndrome,
* Ganglionopathy by Sjögren's syndrome, or paraneoplastic syndrome with Anti- Hu Antibodies, chemotherapy induced (cis-platine, oxaliplatine).
* Positive family history of FAP or FAC
* Proven AL amyloidosis

The new criteria after amendment New eligibility criteria from the 351st patient:

* A. Adults > 50 years old B1. Progressive axonal polyneuropathy

Has:

* Deterioration of EMG sensory potentials >30% in less than 6 months by the same electrophysiology team Where -. Clinical worsening over 6 months, i.e. + 1 ONLS point, or extension of sensory disorders (subjective, objective), or reduction in walking distance, or JAMAR -10% OR B2. Atypical chronic polyradiculoneuritis (CIDP)

  1. with pure sensitive
  2. pure motor
  3. . Asymmetrical sensorimotor impairment predominantly in the upper limbs
  4. Situations C, D, E -even at high protein content on CSF- and as defined by the French group for the study of CIDP C. Peripheral neuropathy evolving for ≥ 12 months and < 10 years. D. Peripheral neuropathy documented by abnormal ENMG (Electroneuromyography).

And

At least one of the following criteria:

1. Chronic polyneuropathy with dysautonomia (orthostatic hypotension)
2. Disabling neuropathy (walking or balance disorders, functional impairment of the hands)
3. Unintentional weight loss of > 5 kg in the last 5 years
4. History of operated carpal tunnel syndrome

Exclusion criteria A. Amyloid deposit characterized by biopsy B. Causes of chronic polyneuropathy: sensory neuropathy typical of diabetes mellitus, chronic alcohol intoxication (women: >14 drinks/week; men >21 drinks/week), vitamin B12 deficiency, chemotherapy (cis-Platin, oxaliplatin) C. CIDP responding to IVIG or corticosteroids (1 point improvement in ONLS) D. Peripheral neuropathy evolving for >10 years E. Dysimmune neuropathy defined by

* with Ac anti-MAG,
* POEMS, CANOMAD,
* Ganglionopathy linked to Gougerot Sjögren's syndrome, to a paraneoplastic syndrome with Anti-Hu antibodies), F. Family history of FAP or FAC (familial amyloid neuropathy or cardiomyopathy) G. AL Amyloidosis

Min Age: 51 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multicentric prospective population in tertiary referal center for neuromuscular diseases
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Rate of amyloidogenic TTR mutation | 1 day
  Rate of amyloidogenic TTR mutation in progressive idiopathic polyneuropathy

SECONDARY OUTCOMES:
To identify the rate of amyloidogenic TTR mutation in different subgroups of patients with neuropathy | 1 day
  Rate of amyloidogenic TTR mutation in different subgroups of patients with neuropathy : disabling neuropathy (including ataxic).
To identify the rate of amyloidogenic TTR mutation in different subgroups of patients with neuropathy :variant Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) | 1 day
  Rate of amyloidogenic TTR mutation in different subgroups of patients with neuropathy :variant Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
To identify the rate of amyloidogenic TTR mutation in different subgroups of patients with neuropathy : upper limb onset neuropathy. | 1 day
  Rate of amyloidogenic TTR mutation in different subgroups of patients with neuropathy : upper limb onset neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: David ADAMS, Principal Investigator — Bicetre Hospital
Locations (10):
- France (10):
  - Chu Bicetre, Le Kremlin-Bicêtre, Kremlin Bicetre
  - CHU Martinique, Martigues, Martinique
  - CHU Saint Etienne, Saint-Etienne, Saint Etienne
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - CHU La Timone, Marseille
  - Hopital guy-de-Chauliac, Montpellier
  - Hôpital de La Salpetrière, Paris
  - Hopital de Hautepierre, Strasbourg